CLINICAL TRIAL: NCT06769568
Title: The Safety and Efficacy of Reduced-dose Conditioning Regimen Containing TBI in Hematopoietic Stem Cell Transplantation Treating Elderly Patients With Aplastic Anemia
Brief Title: Reduced-dose Conditioning Regimen Containing TBI in HSCT Treating Elderly Patients With Aplastic Anemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024078
Record Dates: First submitted 2024-10-23; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Aplastic Anaemia; HSCT; TBI; Old Age
Keywords: aplastic anemia; HSCT; old age; conditioning regimen
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- reduced-dose conditioning regimen containing TBI in hematopoietic stem cell transplantation treating (Experimental): reduced-dose conditioning regimen containing TBI in hematopoietic stem cell transplantation treating elderly patients with aplastic anemia
  Interventions: Drug: reduced-dose conditioning regimen containing TBI in hematopoietic stem cell transplantation treating elderly patients with aplastic anemia

INTERVENTIONS:
Drug: reduced-dose conditioning regimen containing TBI in hematopoietic stem cell transplantation treating elderly patients with aplastic anemia — reduced-dose conditioning regimen containing TBI in hematopoietic stem cell transplantation treating elderly patients with aplastic anemia

SUMMARY:
The TBI-containing reduced-dose conditioning regimen was used to treat elderly patients with aplastic anemia who received hematopoietic stem cell transplantation. The overall survival rate, GVHD-free survival rate, all-cause mortality,et al were studied. The modified conditioning regimen included TBI 2Gy, -7d, busulfan 3.2mg / kg-6d ; fludarabine 30mg / m2 / d-5 ~ -1d ; cyclophosphamide 25-30mg / kg / d-5 ~ -2d ; ATG ( rabbit ) 2 mg / kg / d-5 ~ -1d.

ELIGIBILITY:
Inclusion Criteria:

* ( 1 ) Diagnosis of aplastic anemia, including very severe aplastic anemia, severe aplastic anemia, chronic aplastic anemia and hepatitis-associated aplastic anemia.

( 2 ) Age older than or equal to 50 years old. ( 3 ) Informed consent can be signed by themselves. ( 4 ) HIV negative, HBV, HCV negative. ( 5 ) Informed consent must be signed before the start of the study procedure. Informed consent must be signed by the patient or immediate family members who are 18 years old or older. Considering the patient 's condition, if the patient 's signature is not conducive to the treatment of the disease, the informed consent is signed by the legal guardian or the patient 's immediate family.

Exclusion Criteria:

* ( 1 ) Patients who underwent more than one time of transplantation before enrollment ; ( 2 ) Uncontrolled infection, mechanical ventilation or hemodynamic instability at the time of enrollment ; ( 3 ) Diagnosis of clinically significant severe liver dysfunction ( defined as Child-Pugh C grade ) within 5 days before enrollment ; or within 5 days before enrollment, AST or ALT was 5 times higher than the upper limit of normal, or serum total bilirubin was 2 times higher than the upper limit of normal ; ( 4 ) End-stage renal insufficiency was diagnosed within 5 days before enrollment, and creatinine clearance rate was less than 10ML / min.

( 5 ) Simultaneous diagnosis of moderate hepatic insufficiency and moderate renal insufficiency ( moderate hepatic insufficiency was defined as Child-Pugh B grade ; moderate renal insufficiency was defined as creatinine clearance rate less than 50ML / min ).

( 6 ) In addition to localized basal cell or squamous cell skin cancer or treatment conditions ( such as lymphoma ), there are active solid tumor malignant tumors.

( 7 ) There was active HIV replication before enrollment. HCV antibody positive, HCV-RNA positive, or HBsAg positive could be detected within 90 days before enrollment. The serological response to HIV or active hepatitis C virus is known to be positive.

( 8 ) Having a mental illness or other condition that does not cooperate with the requirements of research, treatment and monitoring.

( 9 ) unable or unwilling to sign the consent form. ( 10 ) Patients with other special conditions who were assessed as unqualified by the researchers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 year after HSCT
  2-year overall survival